CLINICAL TRIAL: NCT04437849
Title: Trial Clínico: Utilidad Del Telemonitoreo en Pacientes Con IC Como Medio de Apoyo Para la autogestión de la Enfermedad
Brief Title: Home Telemonitoring System for Patients With Heart Failure vs Usual Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Tucuman (Other)
Responsible Party: Principal Investigator, Lucía María Yanicelli, Principal Investigator PhD in Exact Sciences and Engineering, Universidad Nacional de Tucuman
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0094
Record Dates: First submitted 2020-06-12; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemonitoring (Experimental)
  Interventions: Device: Home Telemonitoring System
- Usual Care (No Intervention)

INTERVENTIONS:
Device: Home Telemonitoring System — Home Telemonitoring System (HTS) The HTS consists of an App that daily collects measurements of weight, blood pressure, heart rate and symptoms (checklist of symptoms questions). The HTS processes the data and generates and sends an alert to the physicians if a risk situation occurs (measurements are outside of normal ranges). The App has also an educational functionality that allows learning about lifestyle, self-care and healthy habits for HF patients. For this purpose, the application: a) has a section that answers frequent questions, b) has a question and answer game about HF, and c) sends educational messages to the patients every day.
  Arms: Telemonitoring

SUMMARY:
This randomized controlled clinical trial compares a home telemonitoring system (HTS) versus usual care during a 90 days follow-up period of Heart Failure (HF) ambulatory patients, in order to evaluate if the use of the HTS improves quality of life and HF related-knowledge. The study was reviewed and approved by the Methodological Committee and by the Research Ethics Committee from the Provincial Health System, according to the Declaration of Helsinki. Written informed consent was obtained before randomization.

ELIGIBILITY:
Inclusion Criteria:

* were over 18 years with a primary diagnosis of HF,
* had been hospitalized at least once time as a consequence of a HF decompensation,
* had a Smartphone,
* had access to WiFi,
* had access to a weight scale and to a blood-pressure monitor

Exclusion Criteria:

* illiterate patients,
* had learning difficulties,
* had a cognitive impairment sufficient to interfere with the use of the telemonitoring system, or had a severe depression that could interfere with their quality of life perception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Changes in quality of life through the Minnesota Living with Heart Failure Questionnaire (MLHFQ) | 3-month
Changes in HF related knowledge through the Knowledge of CHF questionnaire | 3-month

CONTACTS AND LOCATIONS:
Locations (1):
- Zenón Santillán Health Center Hospital, San Miguel de Tucumán, Tucumán Province, Argentina